CLINICAL TRIAL: NCT04128007
Title: A Phase 2b, 8-Week, Parallel Group, Double Blind, Vehicle-Controlled Study of the Safety and Efficacy of ARQ-154 Foam 0.3% Administered QD in Adolescents and Adults With Scalp and Body Psoriasis
Brief Title: Safety and Efficacy of ARQ-154 Foam in Adolescent and Adult Subjects With Scalp and Body Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARQ-154-204
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Results first posted 2022-09-30 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARQ-154 foam 0.3% (Experimental): active
  Interventions: Drug: Roflumilast foam 0.3%
- ARQ foam VehicleRQ-154 foam Vehicle (Placebo Comparator): placebo
  Interventions: Drug: Vehicle foam

INTERVENTIONS:
Drug: Roflumilast foam 0.3% — experimental
  Other Names: ARQ-154
  Arms: ARQ-154 foam 0.3%
Drug: Vehicle foam — experimental
  Other Names: placebo
  Arms: ARQ foam VehicleRQ-154 foam Vehicle

SUMMARY:
This study will assess the safety and efficacy of ARQ-154 foam vs placebo applied once a day for 56 days by subjects with scalp and body psoriasis

DETAILED DESCRIPTION:
This is a parallel group, double blind, vehicle-controlled study in which ARQ-154 foam or vehicle is applied once daily x 8 weeks to adolescent and adult subjects with scalp and body psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Participants legally competent to read, write, sign and give informed consent, or, in the case of adolscents, assent with consent of a parent(s) or legal guardian, as required by local laws.
* Males and females ages 12 years and older (inclusive) at the time of consent for assent (for adolescents).
* Scalp psoriasis with an Investigator Global Assessment of Scalp disease severity (S-IGA) of at least Mild ('2') at Baseline.
* A Psoriasis Scalp Severity Index (PSSI) score of at least 6 at Baseline.
* A PASI score of at least 2 (excluding the palms and soles) at Baseline.
* Clinical diagnosis of psoriasis vulgaris of at least 6 months duration as determined by the Investigator. Stable disease for the past 4 weeks.
* Females of childbearing potential (FOCBP) must have a negative serum pregnancy test at Screening (Visit 1) and a negative urine pregnancy test at Baseline (Visit 2).
* Females of non-childbearing potential must either be post-menopausal with spontaneous amenorrhea for at least 12 months or have undergone surgical sterilization.
* Subjects in good health as judged by the Investigator, based on medical history, physical examination, vital signs, serum chemistry labs, hematology values, and urinalysis.
* Subjects are considered reliable and capable of adhering to the Protocol and visit schedule according to the Investigator judgment.

Exclusion Criteria:

* Subjects who cannot discontinue medications and treatments prior to the Baseline visit and during the study according to Excluded Medications and Treatments.
* Planned excessive exposure of treated area(s) to either natural or artificial sunlight, tanning bed or other LED.
* Subjects currently taking lithium or antimalarial drugs.
* Planned initiation or changes to concomitant medication that could, in the opinion of the Investigator, affect psoriasis vulgaris (e.g. beta blockers, ACE inhibitors).
* Current diagnosis of non-plaque forms of psoriasis (e.g., guttate, erythrodermic/exfoliative, palmoplantar only involvement, or pustular psoriasis). Current diagnosis of drug-induced psoriasis.
* Subjects with any condition on the treatment area which, in the opinion of the Investigator, could confound efficacy measurements.
* Known allergies to excipients in ARQ-154.
* Subjects who cannot discontinue the use of strong P-450 cytochrome inhibitors e.g., indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, ketoconazole, nefazodone, saquinavir, suboxone and telithromycin for two weeks prior to the Baseline visit (Visit 2) and during the study.
* Subjects who cannot discontinue the use of strong P-450 cytochrome inducers e.g., efavirenz, nevirapine, glucocorticoids, barbiturates (including phenobarbital), phenytoin, rifampin, and carbamazepine for two weeks prior to the Baseline visit (Visit 2) and during the study.
* Subjects with PHQ-8 >/= 10 or modified PHQ-A >/= 10 at Screening or Baseline.
* Females who are pregnant, wishing to become pregnant during the study, or are breast-feeding.
* Subjects with any serious medical condition or laboratory abnormality that would prevent study participation or place the subject at significant risk, as determined by the Investigator.
* Subjects with a history of chronic alcohol or drug abuse within 6 months of initiation of the investigational product.
* Subjects with a history of a major surgery within 4 weeks prior to Baseline (Visit 2) or has a major surgery planned during the study.
* Subjects who are unable to communicate, read or understand the local language, or who display another condition, which in the Investigator's opinion, makes them unsuitable for clinical study participation.
* Current or a history of cancer within 5 years with the exception of fully treated skin basal cell carcinoma, cutaneous squamous cell carcinoma or carcinoma in situ of the cervix.
* Subjects with active infection that required oral or intravenous administration of antibiotics, antifungal, or antiviral agents within 7 days of Baseline/Day 0.
* Subjects who are family members of the clinical study site, clinical study staff, or sponsor, or family members residing in the same household of enrolled subjects.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, MD, Study Director — Arcutis Biotherapeutics
Locations (47):
- United States (31):
  - Arcutis Biotherapeutics Clinical Site 71, Rogers, Arkansas
  - Arcutis Biotherapeutics Clinical Site 72, Fremont, California
  - Arcutis Biotherapeutics Clinical Site 85, San Diego, California
  - Arcutis Biotherapeutics Clinical Site 21, Cromwell, Connecticut
  - Arcutis Biotherapeutics Clinical Site 91, Boynton Beach, Florida
  - Arcutis Biotherapeutics Clinical Site 20, Coral Gables, Florida
  - Arcutis Biotherapeutics Clinical Site 88, Miami, Florida
  - Arcutis Biotherapeutics Clinical Site 90, Miami, Florida
  - Arcutis Biotherapeutics Clinical Site 83, Sweetwater, Florida
  - Arcutis Biotherapeutics Clinical Site 99, Rolling Meadows, Illinois
  - Arcutis Biotherapeutics Clinical Site 78, Indianapolis, Indiana
  - Arcutis Biotherapeutics Clinical Site 95, Plainfield, Indiana
  - Arcutis Biotherapeutics Clinical Site 77, Louisville, Kentucky
  - Arcutis Biotherapeutics Clinical Site 79, Covington, Louisiana
  - Arcutis Biotherapeutics Clinical Site 94, Metairie, Louisiana
  - Arcutis Biotherapeutics Clinical Site 73, Fridley, Minnesota
  - Arcutis Biotherapeutics Clinical Site 84, Saint Joseph, Missouri
  - Arcutis Biotherapeutics Clinical Site 98, Portsmouth, New Hampshire
  - Arcutis Biotherapeutics Clinical Site 87, High Point, North Carolina
  - Arcutis Biotherapeutics Clinical Site 96, Bexley, Ohio
  - Arcutis Biotherapeutics Clinical Site 82, Portland, Oregon
  - Arcutis Biotherapeutics Clinical Site 80, Broomall, Pennsylvania
  - Arcutis Biotherapeutics Clinical Site 97, Murfreesboro, Tennessee
  - Arcutis Biotherapeutics Site 70, Arlington, Texas
  - Arcutis Biotherapeutics Clinical Site 76, Austin, Texas
  - Arcutis Biotherapeutics Clinical Site 86, College Station, Texas
  - Arcutis Biotherapeutics Clinical Site 74, Houston, Texas
  - Arcutis Biotherapeutics Clinical Site 89, Pflugerville, Texas
  - Arcutis Biotherapeutics Clinical Site 93, San Antonio, Texas
  - Arcutis Biotherapeutics Clinical Site 81, Norfolk, Virginia
  - Arcutis Biotherapeutics Clinical Site 75, Richmond, Virginia
- Australia (4):
  - Arcutis Biotherapeutics Clinical Site 51, Kogarah, New South Wales
  - Arcutis Biotherapeutics Clinical Site 52, Westmead, New South Wales
  - Arcutis Biotherapeutics Clinical Site 54, Hectorville, South Australia
  - Arcutis Biotherapeutics Clinical Site 50, East Melbourne, Victoria
- Bulgaria (5):
  - Arcutis Biotherapeutics Clinical Site 11, Pleven
  - Arcutis Biotherapeutics Clinical Site 13, Sevlievo
  - Arcutis Biotherapeutics Clinical Site 14, Sofia
  - Arcutis Biotherapeutics Clinical Site 10, Sofia
  - Arcutis Biotherapeutics Clinical Site 12, Stara Zagora
- Canada (7):
  - Arcutis Biotherapeutics Clinical Site 64, Calgary, Alberta
  - Arcutis Biotherapeutics Clinical Site 61, Barrie, Ontario
  - Arcutis Biotherapeutics Clinical Site 60, London, Ontario
  - Arcutis Biotherapeutics Clinical Site 62, Peterborough, Ontario
  - Arcutis Biotherapeutics Clinical Site 63, Waterloo, Ontario
  - Arcutis Biotherapeutics Clinical Site 66, Montreal, Quebec
  - Arcutis Biotherapeutics Clinical Site 65, Westmount, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Roflumilast Foam 0.3%: Participants applied roflumilast foam 0.3% once daily (QD) for 8 weeks. Areas of application were all areas affected, including the scalp, face, trunk, and intertriginous regions. There was a 1-week follow-up period after completing treatment.
- Vehicle Foam: Participants applied vehicle foam QD for 8 weeks. Areas of application were all areas affected, including the scalp, face, trunk, and intertriginous regions. There was a 1-week follow-up period after completing treatment.
Period: Overall Study
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Started | 200 | 104
Completed | 177 | 87
Not Completed | 23 | 17
Not completed — Withdrawal by Subject | 9 | 6
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 8 | 7
Not completed — Adverse Event | 5 | 2
Not completed — Not reported | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Roflumilast Foam 0.3%: Participants applied roflumilast foam 0.3% QD for 8 weeks. Areas of application were all areas affected, including the scalp, face, trunk, and intertriginous regions. There was a 1-week follow-up period after completing treatment.
- Total: Total of all reporting groups
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam | Total
Number analyzed (Participants) | 200 | 104 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (14.22) | 45.0 (15.76) | 45.1 (14.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 47 | 143
  Male | 104 | 57 | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 25 | 63
  Not Hispanic or Latino | 161 | 79 | 240
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 4 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 9 | 6 | 15
  White | 180 | 91 | 271
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 3 | 1 | 4
Scalp Investigator Global Assessment (S-IGA) Baseline Score [Count of Participants; unit: Participants] — The S-IGA is 5-point scale assessing the severity of plaque psoriasis on the scalp, with scores ranging from 0 ('clear') to 4 ('severe'). Higher scores indicate greater symptom severity. Population: Two participants in the Roflumilast Foam 0.3% arm did not have baseline S-IGA assessments.
  Participants
    0 - clear: number analyzed (Participants) | 198 | 104 | 302
    0 - clear | 0 | 0 | 0
    1 - almost clear: number analyzed (Participants) | 198 | 104 | 302
    1 - almost clear | 0 | 0 | 0
    2 - mild: number analyzed (Participants) | 198 | 104 | 302
    2 - mild | 18 | 14 | 32
    3 - moderate: number analyzed (Participants) | 198 | 104 | 302
    3 - moderate | 151 | 80 | 231
    4 - severe: number analyzed (Participants) | 198 | 104 | 302
    4 - severe | 29 | 10 | 39
Psoriasis Scalp Severity Index (PSSI) Baseline Score [Mean (Standard Deviation); unit: score on a scale] — The PSSI measures the extent of psoriasis involvement and the severity of erythema, induration, and desquamation of the scalp. Involvement and severity of psoriasis for the PSSI is scored using a scale of 0 to 72, where 0 = no psoriasis and higher scores indicate greater symptom severity. Population: Two participants did not have a baseline PSSI assessment.
  score on a scale
    number analyzed (Participants) | 198 | 104 | 302
    (all) | 22.4 (12.52) | 20.9 (11.70) | 21.9 (12.25)
Body Investigator Global Assessment (B-IGA) Baseline Score [Count of Participants; unit: Participants] — The B-IGA is 5-point scale assessing the severity of plaque psoriasis on the body, with scores ranging from 0 ('clear') to 4 ('severe'). Higher scores indicate greater symptom severity. Population: Two participants in the Roflumilast Foam 0.3% arm did not have baseline B-IGA assessments.
  Participants
    0 - clear: number analyzed (Participants) | 198 | 104 | 302
    0 - clear | 0 | 0 | 0
    1 - almost clear: number analyzed (Participants) | 198 | 104 | 302
    1 - almost clear | 0 | 0 | 0
    2 - mild: number analyzed (Participants) | 198 | 104 | 302
    2 - mild | 69 | 39 | 108
    3 - moderate: number analyzed (Participants) | 198 | 104 | 302
    3 - moderate | 119 | 60 | 179
    4 - severe: number analyzed (Participants) | 198 | 104 | 302
    4 - severe | 10 | 5 | 15
Scalp Itch Numeric Rating Scale (SI-NRS) Baseline Score [Mean (Standard Deviation); unit: score on a scale] — The SI-NRS is a simple, single item scale to assess the participant-reported severity of scalp itch, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the participant experienced in the past 24 hours. Higher scores indicate greater symptom severity.
  score on a scale | 6.4 (2.35) | 6.6 (2.25) | 6.5 (2.31)
Psoriasis Symptom Diary (PSD) Total Baseline Score [Mean (Standard Deviation); unit: units on a scale] — The PSD is a 16-item questionnaire asking subjects to rate the severity of psoriasis-related symptoms in the past 24 hours. Each question is scored from 0 ("no symptoms") to 10 ("worst imaginable symptoms"). Scores range from 0 to 160, with higher scores indicating greater symptom severity.
  units on a scale | 78.5 (39.92) | 84.3 (38.76) | 80.5 (39.55)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Success in the Scalp Investigator Global Assessment (S-IGA) Scale
Description: The number of participants achieving success in the S-IGA scale is presented for each arm. Success is defined as an S-IGA score of 0 ('clear') or 1 ('almost clear'), plus a 2-grade improvement from baseline.The S-IGA is 5-point scale assessing the severity of plaque psoriasis on the scalp, with scores ranging from 0 ('clear') to 4 ('severe'). Higher scores indicate greater symptom severity.
Time Frame: Week 8
Population: All randomized participants with S-IGA score at baseline ≥2 and data available are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 181 | 88
Participants | 107 | 10
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; S-IGA Success at Week 8 Odds Ratio; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by country, baseline S-IGA, and baseline B-IGA per randomization with multiple imputation of missing data; Odds Ratio (OR) = 14.65, 95% CI 2-sided [6.64 to 32.32] — Stratified by country, baseline S-IGA, and baseline B-IGA per randomization with multiple imputation of missing data

2. Secondary Outcome: Number of Participants Achieving Body Investigator Global Assessment (B-IGA) Success at Week 8
Description: The number of participants achieving success in the B-IGA scale is presented for each arm. Success is defined as a B-IGA score of 0 ('clear') or 1 ('almost clear'), plus a 2-grade improvement from baseline. The B-IGA is 5-point scale assessing the severity of plaque psoriasis on the body, with scores ranging from 0 ('clear') to 4 ('severe'). Higher scores indicate greater symptom severity.
Time Frame: Week 8
Population: All randomized participants with data available and baseline B-IGA score ≥2 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 181 | 88
Participants | 73 | 6
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; B-IGA Success at Week 8 Odds Ratio; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by country, baseline S-IGA, and baseline B-IGA per randomization with multiple imputation of missing data; Odds Ratio (OR) = 8.80, 95% CI 2-sided [3.65 to 21.18] — Stratified by country, baseline S-IGA, and baseline B-IGA per randomization with multiple imputation of missing data

3. Secondary Outcome: Number of Participants Achieving Success in Scalp Itch Numerical Rating Scale (SI-NRS) Score
Description: The number of participants with a baseline SI-NRS score ≥4 who achieve success (a ≥4-point improvement from Baseline) at Weeks 2, 4, and 8 is presented for each arm. The SI-NRS is a participant-reported rating of severity of itch at its highest intensity during the previous 24-hour period. The scale ranges from 0 ('no itch') to 10 ('worst imaginable itch'), with higher scores indicating greater symptom severity. Results are based on observed data only.
Time Frame: Baseline and Weeks 2, 4, 8
Population: All randomized participants with baseline SI-NRS score ≥4 with data available are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 166 | 90
Participants
  Week 2 | 74 | 14
  Week 4: number analyzed (Participants) | 158 | 86
  Week 4 | 98 | 19
  Week 8: number analyzed (Participants) | 155 | 81
  Week 8 | 110 | 15
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; SI-NRS Success at Week 2 Odds Ratio; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by country, baseline S-IGA, and baseline B-IGA per randomization with multiple imputation of missing data; Odds Ratio (OR) = 4.06, 95% CI 2-sided [2.14 to 7.71] — Stratified by country, baseline S-IGA, and baseline B-IGA per randomization with multiple imputation of missing data
Statistical Analysis 2: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; SI-NRS Success at Week 4 Odds Ratio; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Stratified by country, baseline S-IGA, and baseline B-IGA per randomization with multiple imputation of missing data; Odds Ratio (OR) = 5.36, 95% CI 2-sided [2.93 to 9.78] — Stratified by country, baseline S-IGA, and baseline B-IGA per randomization with multiple imputation of missing data
Statistical Analysis 3: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; SI-NRS Success at Week 8 Odds Ratio; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Stratified by country, baseline S-IGA, and baseline B-IGA per randomization with multiple imputation of missing data; Odds Ratio (OR) = 9.74, 95% CI 2-sided [5.02 to 18.89] — Stratified by country, baseline S-IGA, and baseline B-IGA per randomization with multiple imputation of missing data

4. Secondary Outcome: Change From Baseline in Psoriasis Symptoms Diary (PSD) Score
Description: The change from baseline in total PSD scores at Weeks 4 and 8 is presented for each arm. The PSD is a 16-item questionnaire asking subjects to rate the severity of psoriasis-related symptoms in the past 24 hours. Each question is scored from 0 ("no symptoms") to 10 ("worst imaginable symptoms"). Scores range from 0 to 160, with higher scores indicating greater symptom severity.
Time Frame: Baseline and Weeks 4 and 8
Population: All randomized participants are included, with multiple imputation used for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 200 | 104
score on a scale
  Week 4 | -45.0 [-53.8 to -36.1] | -25.4 [-35.2 to -15.6]
  Week 8 | -55.0 [-64.0 to -46.1] | -27.5 [-37.5 to -17.6]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Comparison of Week 4 Change from Baseline; Test type: Superiority; p < 0.0001, ANCOVA; ANCOVA with country; treatment; and baseline S-IGA, B-IGA, and PSD scores as independent variables with multiple imputation of missing data; Least Squares Mean Difference = -19.6, 95% CI 2-sided [-27.4 to -11.8] — ANCOVA with country; treatment; and baseline S-IGA, B-IGA, and PSD scores as independent variables with multiple imputation of missing data
Statistical Analysis 2: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Comparison of Week 8 Change from Baseline; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 4, analysis 1]; Least Squares Mean Difference = -27.5, 95% CI 2-sided [-35.5 to -19.5] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Time to Achieve a 50% Reduction From Baseline in Psoriasis Scalp Severity Index (PSSI-50) Score
Description: The time to achieve PSSI-50 (i.e., a 50% reduction from baseline in PSSI score) is presented for each arm. The PSSI measures the extent of psoriasis involvement and the severity of erythema, induration, and desquamation of the scalp. Involvement and severity of psoriasis for the PSSI is scored using a scale of 0 to 72, where 0 = no psoriasis and higher scores indicating greater symptom severity. Results are based on observed data only.
Time Frame: Up to 8 weeks
Population: All randomized participants are included.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 200 | 104
days | 28.0 [17.0 to 29.0] | NA [67 to NA] — Median and upper bound of 95% CI were not calculable due to low number of cases.
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Time to PSSI-50 Hazard Ratio; Test type: Superiority; p < 0.0001, Log Rank — Stratified by country, baseline S-IGA, and baseline B-IGA per randomization; Hazard Ratio (HR) = 3.940, 95% CI 2-sided [2.764 to 5.616] — Stratified by country, baseline S-IGA, and baseline B-IGA per randomization

6. Secondary Outcome: Number of Participants Achieving Psoriasis Scalp Severity Index-75 (PSSI-75)
Description: The number of participants achieving a 75% reduction in PSSI score (i.e., PSSI-75) from baseline. The PSSI measures the extent of psoriasis involvement and the severity of erythema, induration, and desquamation of the scalp. Involvement and severity of psoriasis for the PSSI is scored using a scale of 0 to 72, where 0 = no psoriasis and higher scores indicate greater symptom severity. Results are based on observed data only.
Time Frame: Week 8
Population: All randomized participants with data available are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 180 | 87
Participants | 121 | 19
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; PSSI-75 at Week 8 Odds Ratio; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Stratified by country, baseline S-IGA, and baseline B-IGA per randomization with multiple imputation of missing data; Odds Ratio (OR) = 9.46, 95% CI 2-sided [4.81 to 18.61] — Stratified by country, baseline S-IGA, and baseline B-IGA per randomization with multiple imputation of missing data

7. Secondary Outcome: Number of Participants Achieving PSSI-90
Description: The number of participants achieving a 90% reduction from baseline PSSI score (i.e., PSSI-90) is presented for each arm. The PSSI measures the extent of psoriasis involvement and the severity of erythema, induration, and desquamation of the scalp. Involvement and severity of psoriasis for the PSSI is scored using a scale of 0 to 72, where 0 = no psoriasis and higher scores indicate greater symptom severity. Results are based on observed data only.
Time Frame: Baseline and Week 8
Population: All randomized participants with data available are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 180 | 87
Participants | 84 | 3
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; PSSI-90 at Week 8 Odds Ratio; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by country, baseline S-IGA, and baseline B-IGA per randomization with multiple imputation of missing data; Odds Ratio (OR) = 34.45, 95% CI 2-sided [8.49 to 139.77] — Stratified by country, baseline S-IGA, and baseline B-IGA per randomization with multiple imputation of missing data

ADVERSE EVENTS:
Time Frame: Up to 9 weeks
Description: All participants who received ≥1 dose of study intervention are included.
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
All-Cause Mortality (participants affected / at risk) | 0/198 | 0/104
Serious Adverse Events (participants affected / at risk) | 1/198 | 0/104
Other Adverse Events (participants affected / at risk) | 0/198 | 0/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roflumilast Foam 0.3% (N=198) | Vehicle Foam (N=104)
Testicular torsion (Reproductive system and breast disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor is supportive of publishing clinical trial findings. Any form of publication that is derived from this study must be submitted to Arcutis, Inc. for review and approval. The process of coordinating publication efforts is detailed in the Clinical Trial Agreement.

DOCUMENTS (2):
  • Study Protocol (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT04128007/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT04128007/SAP_002.pdf